CLINICAL TRIAL: NCT04785820
Title: A 3-Arm, Randomized, Blinded, Active-Controlled, Phase II Study of RO7121661, a PD1-TIM3 Bispecific Antibody and RO7247669, a PD1-LAG3 Bispecific Antibody, Compared With Nivolumab in Participants With Advanced or Metastatic Squamous Cell Carcinoma of the Esophagus
Brief Title: A Study of Lomvastomig (RO7121661) and Tobemstomig (RO7247669) Compared With Nivolumab in Participants With Advanced or Metastatic Squamous Cell Carcinoma of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP42772; 2020-004606-60 (EudraCT Number)
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Advanced or Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lomvastomig (Experimental)
  Interventions: Drug: Lomvastomig
- Tobemstomig (Experimental)
  Interventions: Drug: Tobemstomig
- Nivolumab (Active Comparator)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Lomvastomig — 2100 milligrams (mg) administered by intravenous (IV) infusion once every 2 weeks on Day 1 of each 14-day cycle.
  Other Names: RO7121661; RG7769; PD1-TIM3 BsAb
  Arms: Lomvastomig
Drug: Tobemstomig — 2100 mg administered by IV infusion once every 2 weeks on Day 1 of each 14-day cycle.
  Other Names: RO7247669; RG6139; PD1-LAG3 BsAb
  Arms: Tobemstomig
Drug: Nivolumab — 240 mg administered by IV infusion once every 2 weeks on Day 1 of each 14-day cycle.
  Other Names: Opdivo®
  Arms: Nivolumab

SUMMARY:
This is a Phase II, randomized, blinded, active-controlled, global, multicenter study designed to evaluate the safety and efficacy of lomvastomig and tobemstomig, compared with nivolumab, in patients with advanced or metastatic esophageal squamous-cell carcinoma (ESCC) refractory or intolerant to fluoropyrimidine- or taxane- and platinum-based regimen.

Following approval of the protocol amendment version 3, recruitment into the lomvastomig arm has been stopped. The decision to stop recruitment for lomvastomig was based on strategic considerations and not based on emerging safety and/or efficacy data. The benefit/risk assessment for lomvastomig remains unchanged.

The study was planned to enroll participants randomized in a 1:1:1 ratio to receive lomvastomig, tobemstomig, or nivolumab. With version 3 of the protocol, recruitment into the lomvastomig arm has stopped, and moving forward, participants will be randomized in a 1:1 ratio to receive either tobemstomig or nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic, histologically confirmed esophageal squamous-cell carcinoma (ESCC)
* Patients who have previously received 1 line of treatment with either a fluoropyrimidine- and platinum- or a taxane- and platinum-based regimen in non-curative intention prior to randomization; or patients who received treatment with a fluoropyrimidine-/taxane- and platinum-based regimen in curative intention and had recurrence or progression within 24 weeks after the last dose of the treatment
* Radiologically measurable disease according to RECIST v1.1. Previously irradiated lesions should not be counted as target lesions unless clearly progressed after the radiotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* A life expectancy of at least (≥)12 weeks
* Tissue samples must be provided for analysis of anti-programmed death ligand-1 (PD-L1) tumor positivity
* Adverse events from any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade ≤1, except alopecia (any grade), vitiligo, endocrinopathy managed with replacement therapy, and Grade 2 peripheral neuropathy
* Adequate cardiovascular, hematological, liver, and renal function
* Serum albumin ≥25 grams per liter (g/L),
* For participants not receiving therapeutic anticoagulation: prothrombin time (PT) and activated partial thromboplastin time ≤1.5 times (×) the upper limit of normal (ULN); for participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP), or a WOCBP who agrees to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods during the treatment period and for at least 5 months after the final dose of study drug and have a negative pregnancy test (blood) within the 7 days prior to randomization.
* A male participant must remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures such as a condom plus an additional contraceptive method and refrain from donating sperm during the treatment period and for at least 5 months after the final dose of study drug

Exclusion Criteria:

* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to any of the components of RO7121661, RO7247669, or nivolumab, including but not limited to, hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with significant malnutrition. Patients whose nutrition has been well controlled for ≥28 days prior to randomization may be enrolled
* Evidence of complete esophageal obstruction not amenable to treatment
* Higher risk of bleeding or fistula caused by esophageal lesions invading adjacent organs (aorta or tracheobronchial tree). Patients with manageable fistula may be included at the Investigator's discretion.
* Symptomatic central nervous system (CNS) metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or without evidence that disease has been clinically stable for ≥14 days prior to randomization
* Active or history of carcinomatous meningitis/leptomeningeal disease
* Asymptomatic CNS primary tumors or metastases if they have requirement for steroids or enzyme inducing anticonvulsants in the last 28 days prior to randomization
* Uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry
* Active second malignancy (with some exceptions)
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders, known autoimmune diseases or immune deficiency, or other diseases with ongoing fibrosis (such as scleroderma, pulmonary fibrosis, emphysema, neurofibromatosis, palmar/plantar fibromatosis, etc.).
* Encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* Significant cardiovascular/cerebrovascular disease within 6 months prior to randomization
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial (including but not limited to tuberculosis [TB] and typical mycobacterial disease), parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with intravenous (IV) antibiotics or hospitalization (relating to the completion of the course of antibiotics, except if for tumor fever) within 28 days prior to randomization
* Known clinically significant liver disease, including alcoholic hepatitis, cirrhosis, and inherited liver disease.
* Major surgical procedure or significant traumatic injury (excluding biopsies) within 28 days prior to randomization, or anticipation of the need for major surgery during the course of the study
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Dementia or altered mental status that would prohibit informed consent
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (expected to occur once monthly or more frequently)
* Active or history of autoimmune disease or immune deficiency
* Positive human immunodeficiency virus (HIV) test at screening
* Positive hepatitis B surface antigen (HBsAg) or positive total hepatitis B core antibody (HBcAb) test at screening
* Positive hepatitis C virus (HCV) antibody test at screening
* Prior cancer therapy with any immunomodulatory agents including checkpoint inhibitors (CPIs; such as anti-PDL1/PD1, anti-CTLA-4, anti-LAG3, anti-TIM3)
* Vaccination with live vaccines within 28 days prior to randomization, or anticipation that a live attenuated vaccine will be required during the study
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to randomization
* Concurrent therapy with any other investigational drug (defined as treatment for which there is currently no regulatory authority approved indication) 28 days or 5 half-lives of the drug (whichever is shorter) prior to randomization
* Treatment with immune-modulating and immune suppressive agents/medication 5 half-lives or 28 days (whichever is shorter) prior to randomization
* Regular immunosuppressive therapy (i.e., for organ transplantation, chronic rheumatologic disease)
* Radiotherapy within the last 28 days before start of study drug treatment is not allowed, with the exception of limited palliative radiotherapy
* Prior treatment with adoptive cell therapies, such as chimeric antigen receptor T cells (CAR-T) therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival, Defined as the Time from Randomization to Death from Any Cause | Up to 3.5 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events, Severity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | Up to 3.5 years
Objective Response Rate (ORR), Defined as the Percentage of Participants with a Complete or Partial Response According to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) | Up to 3.5 years
Disease Control Rate (DCR), Defined as the Percentage of Participants with an Objective Response or Stable Disease According to RECIST v1.1 | Up to 3.5 years
Duration of Response for Participants with ORR, Defined as the Time from the First Occurrence of a Documented Objective Response to Disease Progression According to RECIST v1.1 or Death from any Cause, Whichever Occurs First | Up to 3.5 years
Progression-Free Survival (PFS), Defined as the Time from Randomization to the First Occurrence of Progression as Determined According to RECIST v1.1 or Death from any Cause, Whichever Occurs First | Up to 3.5 years
Percentage of Participants Reporting Clinically Meaningful Improvement in Global Health Status/Quality of Life (GHS/QoL), and Emotional and Social Functioning, Defined as a ≥10-Point Increase from Baseline as Measured by the EORTC QLQ-C30 | Baseline (Day 1 of Cycle 1) and Day 1 of Cycles 4, 7, 10, and then every 6 cycles thereafter (each cycle is 14 days) until treatment discontinuation; and every 3 months during the first year of post-treatment follow-up (up to 3 years)
  EORTC QLQ-C30 = European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30
Percentage of Participants Reporting a Clinically Meaningful Improvement in GHS/QoL, and Emotional and Social Functioning, Defined as a ≥10-Point Increase from Baseline as Measured by the EORTC IL97 Questionnaire | Baseline (Cycle 1 Day 1) and Day 1 of Cycles 2, 3, 5, 6, 8, and 9 (each cycle is 14 days)
  EORTC IL97 = European Organisation for Research and Treatment of Cancer - Item Library 97
Percentage of Participants Reporting a Clinically Meaningful Improvement in Dysphagia, Defined as a ≥10-Point Increase from Baseline as Measured by the EORTC QLQ-OES18 | Baseline (Cycle 1 Day 1) and Day 1 of each subsequent treatment cycle (each cycle is 14 days) until treatment discontinuation; and every 3 months during the first year of post-treatment follow-up (up to 3 years)
  EORTC QLQ-OES18 = European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire for Esophageal Cancer
Serum Concentrations of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Area Under the Time-Serum Concentration Curve (AUC) of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Maximum Serum Concentrations of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Total Clearance of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Volume of Distribution at Steady State of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Terminal Half-Life of Tobemstomig and Nivolumab | Predose and at end of infusion on Day 1 of every treatment cycle and on Day 8 of Cycles 1 and 5 (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Number of Participants with Anti-Drug Antibodies (ADAs) to Tobemstomig or Nivolumab at Baseline and During the Study | Predose at Baseline (Day 1 of Cycle 1) and on Day 1 of Cycles 2, 3, 4, 5, and 7, and then every 3 cycles thereafter (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Change from Baseline in the Number of T-cell Subsets by Phenotype and Activation Status (CD4/CD8 HLA-DR+Ki67+) in the Peripheral Blood | Predose at Baseline (Day 1 of Cycle 1) and on Day 1 of Cycles 2, 3, 5, and 7, and then every 3 cycles thereafter (each cycle is 14 days); and at treatment discontinuation (up to 2 years)
Change from Baseline in the Number of CD8+ T-cells Infiltrating the Tumor Microenvironment | Baseline and Day 1 of Cycle 3 (each cycle is 14 days)
Change from Baseline in the Number of CD8+ T-cells Proliferating (CD8+Ki67+) in the Tumor Microenvironment | Baseline and Day 1 of Cycle 3 (each cycle is 14 days)
Baseline PDL1, CD8+PD1+, CD8+TIM3+, and CD8+LAG3+ Expression in the Tumor Microenvironment | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- Argentina (2):
  - Inst. Alexander Fleming, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Brazil (2):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Czechia (2):
  - Masaryk?v onkologický ústav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
- Denmark (2):
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- France (7):
  - Institut Bergonie, Bordeaux
  - Hopital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Hopital Timone Adultes, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - APHP - Hopital Saint Antoine, Paris
  - ICO Rene Gauducheau, Saint-Herblain
- Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok, Hungary
- Italy (3):
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola, Emilia-Romagna
  - Azienda Sanitaria Universitaria Integrata di Udine - PO Universitario Santa Maria della, Udine, Friuli Venezia Giulia
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - Aga Khan University Hospital, Nairobi
- Poland (4):
  - Centrum Onkologii w Bydgoszczy, Bydgoszcz
  - Szpital Morski im. PCK, Gdynia
  - Krakowski Szpital Specjalistyczny im sw. Jana Paw?a II, Krakow
  - NIO im Marii Sklodowskiej-Curie, Warsaw
- Russia (4):
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Moscow Oblast
  - MEDSI Clinical Hospital on Pyatnitsky Highway, Moscow, Moscow Oblast
  - Group of companies "Medci", Moskva, Moscow Oblast
- Singapore (2):
  - National Cancer Centre, Singapore
  - Curie Oncology, Singapore
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (3):
  - Changhua Christian Hospital, Chang-hua
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist.
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (7):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Dicle Uni Medical Faculty, Diyarbakır
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Ac?badem Altunizade Hastanesi, Istanbul
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
  - Van Yuzuncu Yil University Hospital, Van
- Ukraine (2):
  - Communal Non profit Enterprise Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy
- Nottingham City Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing